CLINICAL TRIAL: NCT01335763
Title: Pharmacist Intervention for Glycemic Control in The Community (The RxING Study)
Brief Title: Pharmacist Intervention for Glycemic Control in The Community
Acronym: RxING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Ross T. Tsuyuki, Professor of Medicine (Cardiology) and Director, EPICORE Centre University of Alberta, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_05128*
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
Keywords: HbA1c; Multicentre before-after design; Glycemic control; Community pharmacists
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin glargine (Other): 10 units at bedtime of insulin glargine will be prescribed to the patients who has HbA1c levels of 7.5-11%. Insulin glargine dose is going to be titrated by increments of 1 unit daily by the patient to achieve a morning fasting glucose of <=5.5mmol/L
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin glargine — 10 units at bedtime of insulin glargine will be prescribed to the patients who has HbA1c levels of 7.5-11%. Insulin glargine dose is going to be titrated by increments of 1 unit daily by the patient to achieve a morning fasting glucose of <=5.5mmol/L
  Other Names: Lantus

SUMMARY:
Background: Approximately 1.9 million Canadians are living with diabetes and this is estimated to increase by 75% over the next few decades. Pharmacists are front line primary healthcare professionals who see patients with diabetes frequently and in Alberta, they have been allowed to prescribe medications and order laboratory tests. As such, pharmacists could systematically identify poorly controlled diabetes patients and provide greater access to diabetes interventions to improve blood sugar control.

Objective: The aim of this study is to determine the effect of a community pharmacist intervention on blood sugar control in individuals with poorly controlled diabetes.

Project description:

100 adults with type 2 diabetes and uncontrolled blood sugar will be defined by the participating pharmacists. Blood sugar control is going to assessed using hemoglobin A1c test (a blood test to measure individual's blood sugar control over the last 3 months). This test requires obtaining a blood spot from the patient which will be obtained by pricking his/her fingertip. Based on the hemoglobin A1c test result the pharmacist will assess the patient's need for insulin glargine, if the patient needs insulin glargine the pharmacist is going to prescribe it for him/her and educate him/her on its use. Patients are going to be followed up closely by the pharmacists for 6 months with regular updates to the patients' family physicians. This multi-centre study should demonstrate pharmacists' ability to improve glycemic control and improve access to care.

DETAILED DESCRIPTION:
BACKGROUND/RATIONALE:

Approximately 1.9 million Canadians are living with diabetes. Estimates are that this number will increase by 75% over the next few decades. Glycemic control in patients with type 2 diabetes mellitus is poor, and poorly controlled patients contribute significantly to the cost of primary health care in Canada. 10% of all acute care hospital admissions in 2006 were attributed to diabetes and its complications.

As type 2 diabetes is a progressive disease, most patients with type 2 diabetes will eventually require insulin. In patients who present with type 2 diabetes and a HbA1C over 9%, insulin can be started immediately, however, historically physicians generally perceive their to be patient difficulties in starting insulin therapy.

INSIGHT demonstrated improved glycemic control with addition of insulin glargine to oral hypoglycemic agents in patients with type 2 diabetes. However, physicians are often reluctant to initiate insulin in these patients. In addition, physicians do not have a system to systematically identify potential candidates for insulin add-on therapy

Pharmacists are front line primary care professionals who see patients with diabetes more frequently than family physicians and as such, could systematically and proactively identify patients with type 2 diabetes with poor glycemic control as a public health approach to chronic disease management. This approach has been used successfully by our group in the past with dyslipidemia and hypertension management involving patients with diabetes.

The scope of practice for pharmacists is changing, with legislation in Alberta (and soon other provinces) allowing pharmacists to prescribe Schedule I medications and order laboratory tests. As such, there is an opportunity to provide greater access, convenience and improved glycemic control by engaging community pharmacists and their patients.

PRIMARY OBJECTIVE: To determine the effect of a community pharmacist prescribing intervention on glycemic control in patients with poorly controlled type 2 diabetes.

SECONDARY OBJECTIVES:

* To determine the effects of pharmacist-directed diabetes care focusing on glycemic control on:

  * patient satisfaction
  * quality of life
  * dosage changes of oral agents
  * persistence on insulin glargine and the end of follow-up
  * hypoglycemic episodes
* To conduct a health economic assessment of the costs and benefits of the intervention

METHODS:

Design: multicentre pragmatic before-after design trial

Setting: Ten community pharmacies in Alberta for recruitment and follow-up, engaging both patients and family physicians

• participating pharmacists will have additional prescribing authorization. For pharmacists not having additional prescribing authorization, we will facilitate their application as done in the rural RxACTION study.

Recruitment: Pharmacists will systematically identify potential candidates by inviting all patients with type 2 diabetes receiving oral hypoglycemic medications to check their HbA1c using a point of care test. HbA1c is going to be measured in the pharmacy. The patient has to sign the first stage consent form in order to get his/her HbA1c measured. After signing the consent form, the patient's HbA1c will be measured using a digital meter which requires a blood spot which will be gained by pricking the patient's fingertip. If the result of HbA1c test is normal the patient will be given his/her result and told to keep up the good work. If the result of HbA1c test is high (7.5-11 %) and the patient meets the other inclusion criteria for the study the patient will be asked if he/she wants to participate in the study. If the patient agrees on participating in the study he/she will be asked to sign the second stage consent form. After signing the consent form the patient will be started on insulin glargine at bedtime and will be taught how to use the insulin pen. If HbA1c is > 11% the patient will be assessed by the study investigators, treatment recommendations will be checked and will be referred to his/her family physician.

Follow-up: Patients will be followed at 2, 4, 8, 14, 20, and 26 weeks to capture adverse events, adherence to the insulin regimen, fasting blood sugars (measured by the patient), insulin dose and titration. HbA1c will be measured at baseline and then at week 14 visit and week 26. Interim telephone follow-up may be performed at the discretion of the pharmacist investigator, however telephone follow-up cannot be used for 2 consecutive visits, nor for week 14 or 26 visits. Fasting glucose will be measured at the discretion of the pharmacist and patients will monitor their blood glucose at home and record in a standard patient diary.

After each follow up study the pharmacists is going to inform the patient's family physician if there were any changes in the patient's treatment regimen and also about the results of any tests conducted.

One year after the final follow up visit, the pharmacy is going to receive a phone call from the study investigators to check if the patient is still taking insulin.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 18 years of age
* Type 2 diabetes for at least 6 months
* Taking 1 or more oral hypoglycemic agents
* Patient attending your community pharmacy where you decided that addition of insulin glargine may be of benefit to the patient
* Baseline HbA1c 7.5 - 11%
* Signed informed consent

Exclusion Criteria:

* Have used, or currently using, Insulin
* History of ketoacidosis
* Pregnant
* Works night shift
* Renal impairment(Serum Creatinine: females ≥ 124 mmol/l, males ≥ 133 mmol/l)
* Clinically unstable
* Unwilling/unable to attend follow up visits
* Unlikely to adhere to study procedures (eg. due to cognitive limitations, severe psychiatric disorder or alcoholism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The change in HbA1c from baseline to week 26 | 6 months
  The change of the patients' HbA1c between the baseline and the 26 week visits

SECONDARY OUTCOMES:
Quality of life and patient satisfaction. | 6 months
  Quality of life and patient satisfaction is going to be measured through using the questionnaires Audit of Diabetes-Dependent Quality of Life (ADDQoL), Diabetes Treatment Satisfaction Questionnaire and Diabetes Treatment Satisfaction Questionnaire change (DTSQ and DTSQc)
Proportion of patients achieving the target HbA1c | 6 months
  Proportion of patients achieving HbA1c of ≤7.0% during follow-up
Type and degree of dosage changes in oral hypoglycemic agents | 6 months
  The type and the degree of changes in the oral hypoglycemic dosing regimen
Persistence on insulin glargine | 6 months
  Percentage of patients still taking insulin at the end of follow-up
Safety | 6 months
  Number of hypoglycemic episodes; symptomatic confirmed and severe (i.e., Requiring the help from a third party), as defined by the CDA guidelines
Health economic evaluation | 6 months
  Cost-effectiveness analyses from a healthcare payor (government) perspective. Costs will include pharmacist training, time spent with patients, pharmaceutical care processes (includes number of face-to-face meetings, time spent with the patient, number and duration of phone calls, number and type of testing per patient, equipment and testing costs, medication costs and out of pocket costs for patients). Clinical benefits will be estimated by modeling the A1C reduction with clinical trials estimates of event reductions

CONTACTS AND LOCATIONS:
Locations (1):
- EPICORE Centre, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Al Hamarneh YN, Sauriol L, Tsuyuki RT. After the diabetes care trial ends, now what? A 1-year follow-up of the RxING study. BMJ Open. 2015 Aug 12;5(8):e008152. doi: 10.1136/bmjopen-2015-008152. PMID 26270946
- [Derived] Al Hamarneh YN, Charrois T, Lewanczuk R, Tsuyuki RT. Pharmacist intervention for glycaemic control in the community (the RxING study). BMJ Open. 2013 Sep 24;3(9):e003154. doi: 10.1136/bmjopen-2013-003154. PMID 24068762